CLINICAL TRIAL: NCT06782503
Title: An Evaluation of a Mind-Body Medicine Training Program for Parole Services Division Staff
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of interest by parole division in continuing training.
Sponsor: The Center for Mind-Body Medicine (Other)
Collaborators: Herbert Simon Family Foundation (Unknown)
Responsible Party: Principal Investigator, Julie K. Staples, Research Director, The Center for Mind-Body Medicine, The Center for Mind-Body Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CMBMIndianaPrisons003
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: Resilience; Empathy; Burnout; Stress; Meditation; Mind-body therapies
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Non-controlled repeated measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mind-Body MedicineTraining/Practicum/Group Consultation Sessions (Other): The only arm is a mind-body medicine training program for parole staff. The training program consists of 3 parts: 1. An initial 4-day training; 2. A 2-day practicum; and 3. Four group consultation sessions. .
  Interventions: Other: Mind-Body Medicine Training Program

INTERVENTIONS:
Other: Mind-Body Medicine Training Program — The 4-day training includes lectures and small group participation. Lecture topics cover information on a variety of mind--body techniques and the small groups allow participants to practice the techniques. The 2-day practicum will teach staff the ways in which they can share the skills they have learned one-on-one with parolees and families of parolees. The practicum lectures will provide a review of the mind-body skills and examples of practical applications. The practicum will also include breakout sessions to allow participants to practice their skills. The four 2-hour group consultation sessions will allow time for the trained staff to share their experiences as they teach these skills to others and ask any questions that may arise. These consultations will support the ongoing sharing of mind-body medicine skills with the parolees and the families of parolees.
  Edit

SUMMARY:
The goal of this study is to evaluate the effectiveness of a mind-body medicine training program on parole services staff. The main questions it aims to answer are:

* Will participation in the training increase resilience; empathy; the belief that one can cope with difficult situations; and decrease symptoms of depression, stress, anxiety, and burnout?
* What is the personal and professional impact of the training program?

Sixty staff members of the Indiana Department of Correction Parole Services Division will do the following:

* Attend an initial 4-day mind-body medicine training. Mind-body techniques taught in the training include: meditation; a breathing exercise; biofeedback; guided imagery; expressing oneself through drawings and writing; movement to reduce stress; and family trees to explore family dynamics.
* Attend a 2-day practicum. The 2-day practicum will teach staff the ways in which they can share the skills they have learned one-on-one with parolees and families of parolees.
* Attend 4 biweekly sessions of 2-hour group consultation sessions. The consultations will support the use of the mind-body skills with the parolees.

Participants will also do the following:

* Fill out standardized questionnaires online before and after the training program in order to measure changes in resilience; empathy; the belief that one can cope with difficult situations; and symptoms of depression, stress, anxiety, and burnout.
* Fill out an additional online questionnaire three months after the consultation sessions to determine how trainees are using the mind-body skills in their work.
* Participate in an online group interview to determine how trainees are using the skills and how the training has affected them personally and professionally.

ELIGIBILITY:
Inclusion Criteria for Mind-Body Medicine Training :

* Being a staff member of the Division of Parole Services
* English Speaking
* Being 18 years of age or older
* Able to fully participate in the training and the small groups included in the training

Exclusion Criteria for Mind-Body Medicine Training:

• None: It is expected that all parole staff will be able to fully participate in the training and the small groups included in the training

Inclusion Criteria for Focus Group Participation :

* Completion of the Mind-Body Medicine Training
* Currently supervising parolees
* Teaching or using mind-body skills with their supervised parolees
* Being 18 years of age or older
* English speaking.

Exclusion Criteria for Focus Group Participation:

• None, as long as the trained staff meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on Resilience assessed using the Connor-Davidson Resilience Scale (CD-RISC) after the 4-day training and 3 months after the last group consultation session | Baseline, after the 4-day training, and 3 months after the last group consultation session
  Resilience will be measured using the Connor-Davidson Resilience Scale (CD-RISC). The CD-RISC consists of 25 questions that are rated on a 5-point scale, with higher scores representing greater resilience.
  Change = (Score after the 4-day training) minus (Baseline score); (Score 3 months after the last group consultation session) minus (Score after the 4-day training); and (Score 3 months after the last group consultation session) minus (Baseline score)

SECONDARY OUTCOMES:
Change from Baseline on Coping Self-efficacy assessed using the Coping Self-Efficacy Scale (CSE scale) after the 4-day training and 3 months after the last group consultation session | Baseline, after the 4-day training, and 3 months after the last group consultation session
  Improvements in self-efficacy will be measured using the Coping Self-Efficacy Scale (CSE scale). The CSE scale consists of 26 items that are rated using an 11-point scale that ranges from "0 = Cannot do at all" to "10 = Certain can do". Higher scores indicate greater levels of coping self-efficacy.
  Change = (Score after the 4-day training) minus (Baseline score); (Score 3 months after the last group consultation session) minus (Score after the 4-day training); and (Score 3 months after the last group consultation session) minus (Baseline score)
Change from Baseline on Empathy will be assessed using the Toronto Empathy Questionnaire (TEQ) after the 4-day training and 3 months after the last group consultation | Baseline, after the 4-day training, and 3 months after the last group consultation session
  Improvements in empathy will be measured using the Toronto Empathy Questionnaire (TEQ). The TEQ scale consists of 16 items that are rated using a 5-point scale that ranges from "0 = never" to "4 = always. Higher scores indicate higher levels of empathy.
  Change = (Score after the 4-day training) minus (Baseline score); (Score 3 months after the last group consultation session) minus (Score after the 4-day training); and (Score 3 months after the last group consultation session) minus (Baseline score)
Change from Baseline on Depression, Anxiety, and Stress using the Depression Anxiety and Stress Scale -21 (DASS-21) after the 4-day training and 3 months after the last group consultation session | Baseline, after the 4-day training, and 3 months after the last group consultation session
  The DASS - 21 consists of 7 questions each to measure the emotional states of depression, anxiety, and stress. Higher scores indicated higher levels of depression, anxiety and stress.
  Change = (Score after the 4-day training) minus (Baseline score); (Score 3 months after the last group consultation session) minus (Score after the 4-day training); and (Score 3 months after the last group consultation session) minus (Baseline score)
Change from Baseline Burnout using the Oldenburg Burnout Inventory (OLBI) after the 4-day training and 3 months after the last group consultation session | Baseline, after the 4-day training, and 3 months after the last group consultation session
  Decreases in burnout will be measured with Oldenburg Burnout Inventory (OLBI). The OLBI consists of 16-items that are rated using a 4-point scale that ranges from "1= strongly agree" to "4 = strongly disagree". There are two subscales: Exhaustion and Disengagement. Higher scores indicated greater levels of burnout.
  Change = (Score after the 4-day training) minus (Baseline score); (Score 3 months after the last group consultation session) minus (Score after the 4-day training); and (Score 3 months after the last group consultation session) minus (Baseline score)

OTHER OUTCOMES:
Focus Group for Parole Staff Who Are Using Mind-Body Skills with Their Supervised Parolees | 3 months after the last consultation group
  Focus group interviews determine will how parole staff have been using what was taught in the mind-body medicine training and how the training has affected them, their work, and their supervision of parolees.

CONTACTS AND LOCATIONS:
Overall Officials: Julie K Staples, PhD, Principal Investigator — The Center for Mind-Body Medicine
Locations (1):
- Indiana Department of Correction, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results in the publication
Supporting Information: Study Protocol
Time Frame: January 2028 - no end date
Access Criteria: Any researcher may request the de-identified IPD from the corresponding author and it will be provided by email.

REFERENCES:
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Demerouti E, Mostert K, Bakker AB. Burnout and work engagement: a thorough investigation of the independency of both constructs. J Occup Health Psychol. 2010 Jul;15(3):209-222. doi: 10.1037/a0019408. PMID 20604629
- [Background] Spreng RN, McKinnon MC, Mar RA, Levine B. The Toronto Empathy Questionnaire: scale development and initial validation of a factor-analytic solution to multiple empathy measures. J Pers Assess. 2009 Jan;91(1):62-71. doi: 10.1080/00223890802484381. PMID 19085285
- [Background] Chesney MA, Neilands TB, Chambers DB, Taylor JM, Folkman S. A validity and reliability study of the coping self-efficacy scale. Br J Health Psychol. 2006 Sep;11(Pt 3):421-37. doi: 10.1348/135910705X53155. PMID 16870053
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- See also: This page describes The Center for Mind-Body Medicine Training Program — https://cmbm.org/work-with-us/training/